CLINICAL TRIAL: NCT00484380
Title: Contribution of the Scanner in the Coronary Evaluation Before Valvular Replacement
Brief Title: The Scanner in the Coronary Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: French Federation of Cardiology (Other)
Responsible Party: Pr Gérard Helft, Hôpital de la Pitié Salpêtrière
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006-04
Record Dates: First submitted 2007-06-06; First posted 2007-06-08 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Valvular Disease; Coronary Stenosis
Keywords: Valvular surgery; Diagnostic accuracy of coronary angiography; Coronary stenosis; Coronary revascularisation
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Coronary scanner — multislice spiral computed tomography coronary angiography

SUMMARY:
Conventional coronary angiography is the recommended procedure in detection of coronary stenosis in patients with heart valve disease referred for surgery.The aim of this prospective study is to assess diagnostic accuracy of multislice spiral computed tomography coronary angiography in patients with heart valve disease referred for surgery.

DETAILED DESCRIPTION:
The diagnostic accuracy of multislice spiral computed tomography coronary angiography in terms of sensitivity, specificity, negative and positive predictive value, the conventional coronary angiography being the gold standard.50 patients scheduled for valve surgery will be screened to conduct an additional multislice spiral computed tomography.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for valve surgery who need a conventional coronary angiography
* Informed Content
* Patients affiliated to the social security system

Exclusion Criteria:

* Instable condition
* Arrhythmia including atrial fibrillation
* Impaired renal function
* Known contrast allergy
* Patients unable to hold an apnea during 20 seconds
* Pregnancy
* Emergency
* People unable to sign the informed content such as major under supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The diagnostic accuracy of coronary scanner (sensitivity, specificity, positive and negative predictive values) in the detection of the coronary stenosis higher than 50%. | a month at the latest after the signature of consent

SECONDARY OUTCOMES:
The diagnostic accuracy of coronary scanner to detect the patients requiring or not a coronary revascularisation in more of the valvular surgery. | a month at the latest after the signature of consent

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Helft, MD, PHD, Principal Investigator — Pitié-Salpêtrière Hospital
Locations (1):
- Pitié Salpêtrière Hospital, Paris, France